CLINICAL TRIAL: NCT01632423
Title: A Study of Lumigan® in Patients With Primary Open Angle Glaucoma (POAG) or Ocular Hypertension (OHT)
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: MAF/AGN/OPH/GLA/025
Record Dates: First submitted 2012-06-25; First posted 2012-07-03 (Estimated); Results first posted 2012-09-21 (Estimated); Last update posted 2012-09-21 (Estimated); Status verified 2012-08

CONDITIONS: Glaucoma, Open-Angle; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- POAG or OHT: Patients with POAG or OHT prescribed Lumigan® (bimatoprost 0.01%) treatment in a dose determined by the physician prior to study entry
  Interventions: Drug: bimatoprost 0.01%

INTERVENTIONS:
Drug: bimatoprost 0.01% — Patients with POAG or OHT prescribed Lumigan® (bimatoprost 0.01%) treatment in a dose determined by the physician prior to study entry

SUMMARY:
This is an observational study of Lumigan® 0.01% (bimatoprost) treatment in clinical practice for patients with Primary Open Angle Glaucoma (POAG) or Ocular Hypertension (OHT).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with primary open angle glaucoma or ocular hypertension
* Prescribed Lumigan®

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with open angle glaucoma or ocular hypertension
Sampling Method: Non-Probability Sample
Enrollment: 10337 (Actual)
Dates: Start 2010-02; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Berlin, Germany

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | POAG or OHT
Started | 10337
Completed | 10091
Not Completed | 246

BASELINE CHARACTERISTICS:
Arm/Group | POAG or OHT
Number analyzed (Participants) | 10337
Age Continuous [Mean (Standard Deviation); unit: Years] | 67.27 (12.33)
Sex/Gender, Customized [Number; unit: Participants]
  Female | 5978
  Male | 4307
  Missing Data | 52

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Intraocular Pressure (IOP)
Description: IOP is a measurement of the fluid pressure inside the eye. A negative change from baseline indicates an improvement.
Time Frame: Baseline, 14 Weeks
Population: All enrolled patients with complete data for this outcome measure
Measure: Median (Inter-Quartile Range); unit: Millimeters of Mercury (mmHg)
Arm/Group | POAG or OHT
Number analyzed (Participants) | 10074
Millimeters of Mercury (mmHg)
  Baseline - Right Eye (N=10062) | 20.0 [17.0 to 23.0]
  Change from Baseline at 14 Wks-Rt Eye (N=10062) | -4.0 [-5.0 to -3.0]
  Baseline - Left Eye (N=10074) | 20.0 [17.0 to 23.0]
  Change from Baseline at 14 Wks-Lft Eye (N=10074) | -4.0 [-5.0 to -3.0]

2. Secondary Outcome: Patient Assessment of Tolerability Using a 4-Point Scale
Description: Patient assessment of tolerability using a 4-point scale (very good, good, moderate, and poor). The number of patients assessed as good and very good combined are reported.
Time Frame: 14 Weeks
Population: All enrolled patients with complete data for this outcome measure
Measure: Number; unit: Participants
Arm/Group | POAG or OHT
Number analyzed (Participants) | 9982
Participants | 9227

3. Secondary Outcome: Physician Assessment of Tolerability Using a 4-Point Scale
Description: Physician assessment of tolerability using a 4-point scale (very good, good, moderate, and poor). The number of patients assessed as good and very good combined are reported.
Time Frame: 14 Weeks
Population: All enrolled patients with complete data for this outcome measure
Measure: Number; unit: Participants
Arm/Group | POAG or OHT
Number analyzed (Participants) | 10062
Participants | 9571

4. Secondary Outcome: Patients Who Discontinued Use of Lumigan® Prior to 14 Weeks
Description: Patients who discontinued Lumigan® prior to 14 weeks was assessed as Yes or No.
Time Frame: 14 Weeks
Population: All enrolled patients with complete data for this outcome measure
Measure: Number; unit: Participants
Arm/Group | POAG or OHT
Number analyzed (Participants) | 9459
Participants | 642

5. Secondary Outcome: Patients Who Will Continue Use of Lumigan® After 14 Weeks
Description: Patients who will continue use of Lumigan® after 14 weeks was assessed as Yes or No.
Time Frame: 14 Weeks
Population: All enrolled patients with complete data for this outcome measure
Measure: Number; unit: Participants
Arm/Group | POAG or OHT
Number analyzed (Participants) | 10008
Participants | 9121

ADVERSE EVENTS:
Arm/Group | POAG or OHT
Serious Adverse Events (participants affected / at risk) | 2/10337
Other Adverse Events (participants affected / at risk) | 0/10337
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | POAG or OHT (N=10337)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.